CLINICAL TRIAL: NCT00192738
Title: Does Telephone Follow-up After Discharge Improve Patients Satisfaction and Decrease Hospitalization
Brief Title: Does Telephone Follow-up Improve Patients Satisfaction
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: ZSA1677CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Congestive Heart Failure; Angina Pectoris; Pneumonia; Urinary Tract Infection
Keywords: telephone,; internal medicine,; readmission,; patients' satisfaction
MeSH Terms: conditions — Heart Failure; Angina Pectoris; Pneumonia; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Several studies have shown the importance of Telephone follow-up in reducing hospital readmissions for heart failure. Therefore, we aimed in this cohort to investigate whether telephone follow-up with patients discharged from the general internal department improves patients' satisfaction, increases compliance to treatment and reduces adverse effects. Patients are recruited from the department of general internal medicine who gave informed consent and could communicate. Patients are interviewed by during hospital stay, one and three months later. This group will be compared with patients that are not interviewd by phone aftert hospital discharge.

ELIGIBILITY:
Inclusion Criteria: Ability to sign informed consent and communicate by phone in Hebrew, Arabic, Russian or English -

Exclusion Criteria:Non of the above

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-04; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaher S. Azzam, MD, Principal Investigator — Rambam Medical Center, Ruth & Bruce Rappaport Faculty of Medicine, Technion; Zaher S Azzam, MD, Principal Investigator — Rambam Medical Center, Ruth & Bruce Rappaport Faculty of Medicine
Locations (1):
- Rambam Medical Center, Haifa, Israel